CLINICAL TRIAL: NCT01168128
Title: PERFormance Enhancement of the Canadian Nutrition Guidelines by a Tailored Implementation Strategy: The PERFECTIS Study
Acronym: PERFECTIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daren K. Heyland (Other)
Collaborators: Ministry of Research, Innovation and Science, Ontario (Other); Canadian Foundation for Dietetic Research (CFDR) (Other)
Responsible Party: Sponsor-Investigator, Daren K. Heyland, Director of Clinical Evaluation Research Unit, Clinical Evaluation Research Unit at Kingston General Hospital
Organization: Clinical Evaluation Research Unit at Kingston General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: PERFECTIS
Record Dates: First submitted 2010-07-21; First posted 2010-07-23 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Critically Ill; Intensive Care Unit
Keywords: Enteral Nutrition; Parenteral Nutrition; Critically ill; Nutrition Therapy; Nutrition Support; Practice Guidelines as Topic; Guideline Adherence; Quality Assurance, Health Care; Nutrition Surveys; Questionnaires
MeSH Terms: conditions — Critical Illness; Hyperphagia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tailored Action Plan (Experimental): A Tailored Action Plan is an intervention selected to overcome barriers identified before the design and delivery of the intervention.
  Interventions: Other: Tailored Change Strategy

INTERVENTIONS:
Other: Tailored Change Strategy — e.g. Education, decision support tools

SUMMARY:
Canadian Critical Care Nutrition Guidelines assist health practitioners in identifying best practices for feeding critically ill patients. However, guidelines have resulted in little change in Intensive Care Unit (ICU) practices, possibly because barriers to change differ between ICUs. Change may be facilitated if strategies specifically address identified barriers. The investigators hypothesize that barriers are inversely related to nutrition performance. Tailoring change strategies to overcome barriers to change will reduce the presence of these barriers and lead to improvements in nutrition practice.

DETAILED DESCRIPTION:
A before-after study will be conducted in 7 Canadian and US ICUs. Each participating ICU will implement a tailored guideline implementation intervention aimed at narrowing the guideline-practice gap. The tailored implementation will consist of 4 phases:

1. Audit of Nutrition Practices: The nutrition practice audit will be conducted as part of the data collection for our ongoing international nutrition quality improvement project. This involves collecting data on personal characteristics and nutrition therapy in a consecutive cohort of 20 mechanically-ventilated critically ill adult patients. Performance at each ICU will be assessed by a benchmarked report comparing the nutrition practices to individual recommendations of the Canadian Critical Care Nutrition CPGs, thus enabling identification of the ICUs strengths and weaknesses, and highlighting areas to target for improvement.
2. Barriers Questionnaire: The barriers and enablers questionnaire will be completed by all physicians, all ICU leadership, the dietitian(s), and a random sample of 30 full- and part-time nurses. This questionnaire asks questions about barriers associated with guideline implementation, such as the characteristics of the guidelines, the care provider, the patient, and the context.
3. Tailored Action Plan: Results of the audit of nutrition practices and barriers questionnaire will be evaluated by the investigators and representatives from the Canadian Critical Care Nutrition CPGs Committee. Committee members include research personnel, intensivists, ICU nurse educators, dietitians, and experts in knowledge translation and health services research. They will be responsible for reviewing the benchmarked reports for each participating ICU, identifying the gaps between the key guideline recommendations and what is actually happening in practice, and reviewing the results of the barriers questionnaire to identify the barriers associated with adhering to these specific recommendations at each site. In collaboration with the local opinion leaders, a tailored 12 month action plan will be developed for each individual ICU.

   The specific behavioral change strategies to be implemented as part of the tailored action plan will likely include powerpoint presentations and handouts, packages of key journal articles, reminders (e.g. posters, checklists), system tools (e.g. pre-printed orders, bedside algorithms), interactive web-based tutorials, guidelines on establishing local implementation teams and creating a culture of team work. Prior to the implementation of these behavioral change strategies in the context of the before-after study, focus groups will be conducted to elicit feedback, and revisions made accordingly.
4. Audit of Nutrition Practices: The audit of nutrition practices will be repeated following the 12 month implementation period in order to evaluate changes in nutrition practices.

ELIGIBILITY:
Inclusion Criteria:

* ICUs must be affiliated with a registered dietitian.
* ICUs must have a minimum of 8 beds.
* ICUs must be located in Canada, Australia, or US.
* ICUs have previously participated in the International Nutrition Survey.

Exclusion Criteria:

* ICUs with less than 8 beds.
* ICUs with high nutrition performance, as demonstrated previously in the International Nutrition Survey (i.e. average nutritional adequacy >60% and/or above 50th percentile when ranked against all participating ICUs according to nutrition practice performance score)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2009-09-16 (Actual); Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Feasibility of the study design and intervention | 12 months post implementation of intervention
  Assessed by rate of completion of barriers questionnaires, development of unique tailored action plans at each site, compliance and satisfaction with the tailored action plans, and other user feedback.

SECONDARY OUTCOMES:
Change in nutrition performance score | 20-24 months
  The nutrition performance score is a composite measure including use, timing and adequacy of nutrition, use of small bowel feeds and motility agents, and hyperglycemia. Nutrition performance scores will be calculated after each of the two nutrition practice audits.
Change in barriers to implementation of critical care nutrition clinical practice guidelines | 12 months post implementation of intervention
  Barriers questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Daren K Heyland, MD, Principal Investigator — Clinical Evaluation Research Unit; Heather Stuart, PhD, Principal Investigator — Queen's University; Naomi E Cahill, RD, MSc, Principal Investigator — Queen's University, Clinical Evaluation Research Unit
Locations (5):
- United States (2):
  - Anne Arundel Medical Center, Annapolis, Maryland
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
- Canada (3):
  - Peter Lougheed, Calgary, Alberta
  - Capital Health - University of Alberta Hospital (hospital general systems), Edmonton, Alberta
  - Southlake Regional Health Centre, Newmarket, Ontario

REFERENCES:
- [Background] Jones NE, Dhaliwal R, Day AG, Ouellette-Kuntz H, Heyland DK. Factors predicting adherence to the Canadian Clinical Practice Guidelines for nutrition support in mechanically ventilated, critically ill adult patients. J Crit Care. 2008 Sep;23(3):301-7. doi: 10.1016/j.jcrc.2007.08.004. Epub 2007 Dec 11. PMID 18725033
- [Background] Jones NE, Suurdt J, Ouelette-Kuntz H, Heyland DK. Implementation of the Canadian Clinical Practice Guidelines for Nutrition Support: a multiple case study of barriers and enablers. Nutr Clin Pract. 2007 Aug;22(4):449-57. doi: 10.1177/0115426507022004449. PMID 17644700
- [Background] Cahill NE, Heyland DK. Bridging the guideline-practice gap in critical care nutrition: a review of guideline implementation studies. JPEN J Parenter Enteral Nutr. 2010 Nov-Dec;34(6):653-9. doi: 10.1177/0148607110361907. PMID 21097765
- [Background] Cahill NE, Suurdt J, Ouellette-Kuntz H, Heyland DK. Understanding adherence to guidelines in the intensive care unit: development of a comprehensive framework. JPEN J Parenter Enteral Nutr. 2010 Nov-Dec;34(6):616-24. doi: 10.1177/0148607110361904. PMID 21097762
- [Derived] Cahill NE, Murch L, Cook D, Heyland DK; Canadian Critical Care Trials Group. Implementing a multifaceted tailored intervention to improve nutrition adequacy in critically ill patients: results of a multicenter feasibility study. Crit Care. 2014 May 11;18(3):R96. doi: 10.1186/cc13867. PMID 24887445
- [Derived] Cahill NE, Murch L, Cook D, Heyland DK; Canadian Critical Care Trials Group. Barriers to feeding critically ill patients: a multicenter survey of critical care nurses. J Crit Care. 2012 Dec;27(6):727-34. doi: 10.1016/j.jcrc.2012.07.006. Epub 2012 Sep 13. PMID 22981532
- See also: Clinical Evaluation Research Unit's Critical Care Nutrition website — http://www.criticalcarenutrition.com